CLINICAL TRIAL: NCT06214000
Title: Primary Care-Based Follow-up of Cancer Survivors of the Prostate and Kidney: A Retrospective Study
Brief Title: Primary Care-Based Follow-up of Cancer Survivors of the Prostate and Kidney
Acronym: LiVHOU
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8500
Record Dates: First submitted 2023-12-11; First posted 2024-01-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer; Kidney Cancer
Keywords: Prostate Cancer; kidney cancer
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, the second cancer plan of 2009-2013 aimed to strengthen the role of MT by putting it back at the center of patient monitoring, in particular by asking "regional health agencies to encourage and support local experiments" which aim for better coordination between the city and the hospital. The third cancer plan for 2014-2019 insists on this measure because it had proven to be unproductive, and recommends, in addition to the creation of a nurse dedicated to the coordination of care between community medicine and the hospital, the creation of a direct telephone line to reach the hospital medical team. This measure is mainly aimed at the follow-up of certain cancers that do not require the technical support of the hospital, as is the case in the post-operative follow-up of RCC and CaP, where the additional examinations carried out during follow-up are carried out in the city.

The research hypothesis is that this new method of monitoring had a positive impact on care in terms of quality, accessibility, organization and costs.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old)
* Patient operated on for localized prostate or kidney cancer
* Patient followed at the HUS during the period from 01/01/2015 to 12/31/2021
* Subject who has not expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Patient under active therapy (hormonotherapy, systemic treatment) for the pathology studied
* Impossibility of providing the subject with informed information (difficulties in understanding the subject, etc.)
* Subject under judicial protection
* Subjects under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥18 years old) operated on for localized prostate or kidney cancer during the period from 01/01/2015 to 12/31/2021
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of the economic impact of the treatment of patients operated on for localized prostate or kidney cancer | The period concerned is from January 1, 2015 to December 31, 2021.
  This study concerns a retrospective evaluation of the economic cost of treatment of localized prostate or kidney cancer in patients followed at the University Hospitals of Strasbourg during the period from January 1, 2015 to December 31, 2021.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urologie - CHU de Strasbourg - France, Strasbourg, France